CLINICAL TRIAL: NCT05141786
Title: An Open-label, Multi-center, Non-randomized Phase II Clinical Study to Evaluate the Efficacy and Safety of MRG002 in Patients With HER2-mutated Unresectable/Metastatic Non-small Cell Lung Cancer (NSCLC).
Brief Title: A Study of MRG002 in the Treatment of Patients With HER2-mutated Unresectable/Metastatic Non-small Cell Lung Cancer (NSCLC).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-008
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Non-small- Cell Lung Cancer (NSCLC)
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Non-small-cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002 (Experimental): MRG002 will be administrated via intravenous infusion of 2.6 mg/kg once on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 in patients with HER2-mutated unresectable or metastatic non-small-cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
The trial consists of two stages: efficacy exploration and efficacy verification.

At the first stage, at most 30 patients will be enrolled for each of the two cohorts as defined by HER2 mutation sites. If ≥8 patients achieved objective response, the second stage will be continued; otherwise the trial will be terminated. Approximately 40 patients will be enrolled in the second stage.

ELIGIBILITY:
Inclusion Criteria:

1. Understands and provides written informed consent and willing to follow the requirements specified in protocol.
2. Aged 18 to 75 (including 18 and 75), both genders;
3. Life expectancy ≥ 3 months;
4. Advanced NSCLC patients with HER2 mutation in tumor tissue/blood confirmed by NGS/PCR methods. If no prior test results, a tumor tissue specimen from the most recent archival or biopsy (if archival tissue is not available or sufficient) should be provided.
5. Histologically and/or cytologically confirmed unresectable locally advanced or NSCLC with histological subtype of either non-squamous cell carcinoma or squamous cell carcinoma, and patients have at least one measurable lesion as defined by RECIST v1.1.
6. Patients who have failed at least one prior line of Stand of Care (SOC) therapy. Those who refuse or cannot tolerate chemotherapy can also be enrolled.
7. The score of ECOG for performance status is 0 or 1 with no deterioration within 2 weeks prior to the first dose of the study drug.
8. Radiographic evidence of tumor progression during or after the most recent therapy confirmed by investigator.
9. Organ functions must meet the basic requirements.
10. A negative serum or urine pregnancy test within 72 hours of receiving the first dose of study treatment. A serum pregnancy test is required if the urine pregnancy test is positive or cannot be confirmed negative. Women who are pregnant or breast feeding should be excluded.
11. Adequate contraception for women of childbearing potential is defined as hormonal birth control or an intrauterine device and willingness to use 2 methods of contraception or be surgically sterile, or abstain from hetero sexual activity for the course of the study through 120 days after receiving the last dose of study medications.
12. Male patients must be willing to use a latex condom during any sexual contact with females of childbearing potential during and for 120 days after the last infusion of MRG002, even after having undergone a successful vasectomy.

Exclusion Criteria:

1. Prior treatment with HER2-targeted ADC or HER2 targeted antibody.
2. Histologically/cytologically confirmed small-cell lung cancer (SCLC) and mixed type of lung cancer with SCLC histopathology.
3. Received systemic cytotoxic chemotherapy, small molecule targeted drugs within 3 weeks before the first dose of the study drug; received anti-tumor biological therapy, immunotherapy or major surgery within 4 weeks before first dose of the study drug. Use of any other type of anti-cancer therapy is prohibited throughout the study.
4. Known active CNS metastases and/or carcinomatous meningitis.
5. Presence of severe cardiac dysfunction within 6 months of enrollment.
6. Pulmonary embolism or deep venous thrombosis within 3 months prior to the first dose of the study drug.
7. Known history of malignancy except if the patient has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.
8. Uncontrolled or poorly controlled hypertension. Patients with active bleeding, history of coagulation disorder, or on Coumarin anticoagulant.
9. Known allergic reactions to any component or excipient of MRG002, or known allergic reaction to other prior anti-HER2 (including investigational) or to other monoclonal antibodies ≥ Grade 3.
10. Known active infection, including hepatitis B, hepatitis C. Presence of other significant liver disease.
11. Concurrent, serious, uncontrolled infection or known infection with human immunodeficiency virus (HIV), or have a diagnosed acquired immunodeficiency syndrome (AIDS); or an uncontrolled autoimmune diseases; or previously undergone allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or has previously received a solid organ transplantation.
12. Active uncontrolled bacterial, viral, fungal, rickettsial, or parasitic infection and has not received systemic antibiotics within 14 days unless treated and resolved prior to study treatment.
13. Received a live-viral vaccination within 30 days prior to the first dose of the study drug. Seasonal influenza or approved COVID-19 vaccines that do not contain live virus are allowed.
14. History of moderate to severe dyspnea at rest due to advanced cancer or their complications, severe primary lung disease, current need for continuous oxygen therapy, or any history of interstitial lung disease or pneumonia that required oral or intravenous glucocorticoids to assist with management.
15. Patients who are receiving immunologically based therapy for any reason.
16. History or current active or chronic autoimmune disease, or glomerulonephritis that has required systemic therapy in the past 2 years or who are receiving systemic therapy for an autoimmune or inflammatory disease.
17. Has a clinically significant cardiac condition.
18. Uncontrolled pleural effusion, pericardial effusion, or recurrent ascites requiring ≥ 1 drainage per month.
19. Use of strong CYP3A4 inhibitors or inducers with MRG002 is prohibited due to increased risk of adverse reactions or potential adverse reduction in potential efficacy.
20. Any other disease or clinically significant abnormality in laboratory parameters, or serious medical or psychiatric illnesses/conditions, substance abuse disorder including alcoholism, which in the judgment of the Investigator might compromise the safety of the patient, integrity of the study, interfere with the patient participation in the study, or confound or compromise the study objectives and their interpretability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee (IRC) | Baseline to study completion (up to 12 months).
  ORR is defined as the proportion of subjects with complete response (CR) and partial response (PR) assessed by IRC according to RECIST v1.1.

SECONDARY OUTCOMES:
ORR by Investigator | Baseline to study completion (up to 12 months)
  ORR is defined as the proportion of subjects with CR and PR assessed by investigator according to RECIST v1.1.
Disease Control Rate (DCR) | Baseline to study completion (up to 12 months).
  DCR is defined as the proportion of subjects achieving CR, PR, and stable disease (SD) after treatment.
Duration of Response (DOR) | Baseline to study completion (up to 12 months).
  DOR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Progression Free Survival (PFS) | Baseline to study completion (up to 12 months).
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion (up to 12 months).
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 45 days after the last dose of study treatment.
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
PK parameters: concentration-time curve | Baseline to 30 days after the last dose of study treatment.
  Plot of drug concentration changing with time after drug administration.
Immunogenicity (ADA) | Baseline to 30 days after the last dose of study treatment.
  The proportion of patients with positive ADA results.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No